CLINICAL TRIAL: NCT05352386
Title: Coronary and Heart Effects of Early Treatment in Familial Hypercholesterolemia
Acronym: CHEETAH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: Dutch Heart Foundation (Other)
Responsible Party: Principal Investigator, E.S.stroes, Prof. dr. E.S.G.Stroes, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: NL79640.018.21
Record Dates: First submitted 2022-04-22; First posted 2022-04-28 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-03

CONDITIONS: Familial Hypercholesterolemia
MeSH Terms: conditions — Hyperlipoproteinemia Type II

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Patients with familial hypercholesterolemia, early treated (Other)
  Interventions: Diagnostic Test: Coronary computed tomography angiography (CCTA)
- Patients without familial hypercholesterolemia, late treated (Other)
  Interventions: Diagnostic Test: Coronary computed tomography angiography (CCTA)
- Healthy individuals (Other)
  Interventions: Diagnostic Test: Coronary computed tomography angiography (CCTA)

INTERVENTIONS:
Diagnostic Test: Coronary computed tomography angiography (CCTA) — Participants undergo coronary computed tomography angiography (CCTA)

SUMMARY:
This study evaluates plaque burden and characteristics in early-treated FH patients compared to late-treated FH patients and healthy individuals.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with heterozygous familial hypercholesterolemia or non FH-control
* Adult patients between 25 and 55 years old.

Exclusion Criteria:

* Renal insufficiency, defined as eGFR < 30 ml/min
* Atrial fibrillation
* Any other treatment or clinically relevant condition that could interfere with the conduct or interpretation of the study in the opinion of the investigator
* Inability or unwillingness to comply with the protocol requirements, or deemed by investigator to be unfit for the study.

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 135 (Actual)
Dates: Start 2022-03-07 (Actual); Primary Completion 2022-12-19 (Actual); Study Completion 2022-12-19 (Actual)

PRIMARY OUTCOMES:
Total coronary plaque volume (mm3) | Day 0
Total coronary plaque burden (%) | Day 0

SECONDARY OUTCOMES:
Presence of >50% obstructive stenosis per vessel | Day 0
Presence of <50% nonobstructive stenosis per vessel | Day 0
Calcified coronary plaque volume (mm^3) | Day 0
Calcified coronary plaque burden (%) | Day 0
Non-calcified plaque volume (mm^3) | Day 0
Non-calcified plaque burden (%) | Day 0
Low attenuation plaque volume (mm^3) | Day 0
Low attenuation plaque burden (%) | Day 0
Number of high risk plaque features (positive remodeling, low attenuation plaque, spotty calcification and napkin ring sign) | Day 0
Pericoronary adipose tissue attenuation (Hounsfield units) | Day 0
Plasma LDL cholesterol (mmol/l) | Day 0
Plasma apolipoprotein B (g/l) | Day 0

CONTACTS AND LOCATIONS:
Locations (1):
- Amsterdam UMC, location AMC, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No